CLINICAL TRIAL: NCT05738265
Title: Fluid Resuscitation In Trauma: What Are The Best Strategies And Fluids?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Ragab Ali Ismail, Assistant lacturer, Assiut University
Other Study IDs: FRIT
Record Dates: First submitted 2023-02-01; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- Shocked patients who take crystalloids: Impact of crystalloids on shocked patients in trauma
- Shocked patients who take colloids: Impact of colloids on shocked patients in trauma

SUMMARY:
Illustration of the differential effects of commonly used resuscitation fluids, including isotonic crystalloids, natural and artificial colloids, hypertonic and hyperoncotic solutions to prevent the cellular injury through wiser resuscitation in traumatic patient . The ideal resuscitation strategy for multiply injured patients.

DETAILED DESCRIPTION:
The repletion of patients' intravascular volume through the use of an intravenous (IV) electrolyte solution was first described by a young Irish physician, William Brooke O'Shaughnessy, in 1831. Immersing himself in the middle of a cholera outbreak in Sutherland, England, O'Shaughnessy observed that large amounts of water, sodium, chloride, and bicarbonate were being lost in these patients' stool. With only brain injury as a larger cause of overall mortality, hemorrhage is the leading cause of preventable trauma death. Rates of mortality in injured patients requiring a massive blood transfusion in the late 1980s were greater than 80%. Prehospital strategies considered standard of care at the time included early intravenous (IV) access with 2 large-bore cannulas and aggressive administration of crystalloid, regardless of patient physiology. Most hemorrhage-related deaths occur in the first 6 h after injury The most common reason given for administering resuscitation fluid was impaired tissue perfusion or low measured cardiac output. The next most common indication, was abnormal vital signs (blood pressure, heart rate, urine output or central venous pressure) in the absence of evidence of impaired tissue perfusion Fluids have classically been categorized as crystalloid or colloid, terms introduced by Thomas Graham (Professor of Chemistry, University College London, 1836-1855) long before intravenous fluids were widely used in clinical practice. The ideal fluids should provide a solution to the various components of the physiopathology of shock. Two strategies were proposed to avoid clot disruption and dilutional coagulopathy: delayed resuscitation strategy where fluid is given after bleeding is controlled and permissive hypotension strategy, where fluid is given to increase in systolic blood pressure without reaching normotension. In penetrating trauma patients with hypotension (prehospital Systolic blood pressure < 90 mmHg), delayed resuscitation shows better survival rates compared to immediate resuscitation THE BALANCED RESUSCITATION STRATEGY Ideally, this process begins in the prehospital setting, continues through early trauma bay/emergency room resuscitation, and is completed in the operating room or the ICU, as needed. To improve outcomes of patients undergoing an abbreviated laparotomy or other procedure because of grossly disturbed physiology. As an adjunct to the care of these critically injured patients, its early implementation focused on delivering higher ratios of plasma and platelets, along with other strategies to prevent "popping the clot." Its 3 basic tenets are permissive hypotension, minimizing the use of crystalloid before surgical control of bleeding, and transfusion of blood products in a ratio approximating whole blood

ELIGIBILITY:
Inclusion Criteria:

* The present study will be conducted on shocked patients with multiple trauma of both genders and had 12 years old or more.

Exclusion Criteria:

* patients who are less than 12 years old,haemodynamically stable or with end stage chronic disease . Furthermore ,patients refusing study will be excluded.

Ages: 12 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Impact of resuscitation fluid (crystalloid,colloids) on shocked patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Haemodynamic stability | 1day
  Make the shocked patient haemodynamically stable , systolic blood pressure >90

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelatif, Principal Investigator — Assiut University; Asmaa Elkafafy, Principal Investigator — Alexandria University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Not decided till now

REFERENCES:
- [Result] Finfer S, Liu B, Taylor C, Bellomo R, Billot L, Cook D, Du B, McArthur C, Myburgh J; SAFE TRIPS Investigators. Resuscitation fluid use in critically ill adults: an international cross-sectional study in 391 intensive care units. Crit Care. 2010;14(5):R185. doi: 10.1186/cc9293. Epub 2010 Oct 15. PMID 20950434
- [Result] Shackford SR, Mackersie RC, Holbrook TL, Davis JW, Hollingsworth-Fridlund P, Hoyt DB, Wolf PL. The epidemiology of traumatic death. A population-based analysis. Arch Surg. 1993 May;128(5):571-5. doi: 10.1001/archsurg.1993.01420170107016. PMID 8489391